CLINICAL TRIAL: NCT04407923
Title: Drug Management of Juvenile Idiopathic Arthritis in Covid-19 Context
Brief Title: Drug Management of Juvenile Idiopathic Arthritis in Covid-19 Context : Impact on Therapeutical Managment
Acronym: RHUMAJICOVID
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: RHUMAJICOVID (29BRC20.0148)
Record Dates: First submitted 2020-05-28; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Juvenile Idiopathic Arthritis; COVID 19; Treatment
MeSH Terms: conditions — Arthritis, Juvenile; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current situation of Sars-Cov-2 pandemic generates fears in the general population. Among patients receiving long-term immunomodulatory drugs, especially in the context of auto-immune diseases, there may be legitimates interrogations about the appropriateness of continuing treatment, without modification, in the current context. Juvenile Idiopathic Arthritis is concerns by these fears (the patient and their parents). Patients are treated by several classes of immunomodulatory drugs, including non-steroidal anti-inflammatory drugs, corticosteroids and disease modifying anti-rheumatic drugs. The present study will characterize this issue by defining the proportion of patients whose usual treatment of Juvenile Idiopathic Arthritis has been modified in relation to the actual sanitary crisis, and also to return to school.

ELIGIBILITY:
Inclusion Criteria:

* Juvenile Idiopathic Arthritis satisfying Edmonton criteria
* Ongoing DMARD therapy or AINS for 3 months

Exclusion Criteria:

* Inhability to consent

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Juvenile Idiopathic Arthritis patients with ongoing DMARD therapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-05-25 (Actual); Primary Completion 2020-11-25 (Estimated); Study Completion 2020-11-25 (Estimated)

PRIMARY OUTCOMES:
Reduction or discontinuation of the DMARD therapy in relation to the Covid-19 sanitary crisis | 1 Day
  Reduction or discontinuation of treatment with sDMARD, bDMARD or tsDMARD

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - CH de Belfort, Belfort
  - CHU de Bordeaux, Bordeaux
  - CHRU de Brest, Brest
  - AP-HP Hôpital Kremlin-Bicêtre, Le Kremlin-Bicêtre
  - CHU de Poitiers, Poitiers
  - CHU de Rennes, Rennes
  - CHU de Strasbourg, Strasbourg
  - CHU de Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will be available beginning six months and ending five years following the end study
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.